CLINICAL TRIAL: NCT03574246
Title: The Effect Of Two Packing Types For Throat Pain And Postoperative Nausea And Vomiting During Maxillofacial Surgery
Brief Title: Effects of Two Packing Type in Maxillofacial Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagil Vural, Specialist, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36290600/127
Record Dates: First submitted 2018-05-24; First posted 2018-06-29 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Sore Throat; Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Pharyngitis; Postoperative Nausea and Vomiting | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHXBNZ (Experimental): Pharyngeal pack moisturized with chlorhexidine gluconate %0,12 benzydamine hydrochloride %0,15 and placed to oropharynx
  Interventions: Drug: chlorhexidine gluconate %0,12 benzydamine hydrochloride %0,15
- SF (Active Comparator): Pharyngeal pack moisturized with %0,9 NaCl and placed to oropharynx
  Interventions: Other: %0.9 NaCl Solution

INTERVENTIONS:
Drug: chlorhexidine gluconate %0,12 benzydamine hydrochloride %0,15 — chlorhexidine gluconate + benzydamine hydrochloride oral rinse
  Arms: CHXBNZ
Other: %0.9 NaCl Solution — isotonic sodium chloride
  Arms: SF

SUMMARY:
Operations of oral maxillofacial surgery cause the blood escape into stomach and trachea. Therefore, throat packing is applied. Endotracheal tube cuff is not protective from aspiration. While packing is preventing blood leakage, it may cause postoperative pain due to the pressure. Packing placed between oropharynx and hypopharynx before surgery to prevent leakage to stomach and trachea. The aim of this study is to compare the efficacy of two packing types in throat pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent oral maxillofacial surgery (maxillary and mandibular cysts, orthognathic surgery, palate and alveolar clefts, mandibular and maxillary fractures and reconstruction surgeries) under general anesthesia between the ages of 18-60
2. ASA 1-2 groups of patients
3. Patients who have completed growth and development
4. Patients who are willing to comply with the requirements of the study
5. Patients with complete medical records
6. Operations expected to last at least 2 hours

Exclusion Criteria:

1. Patients with severe systemic disease other than ASA 1-2
2. Difficult entubation story
3. Patients with BMI> 35 kg / m2
4. Contraindications for the use of NSAIDs
5. Patients with diclofenac sodium and metoclopramide allergy
6. Patients whose medical records are inadequate
7. Patients with major tranquilizer or opiate addiction
8. Patients with mental and physical anxiety that would interfere with cooperative operation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperatively 2nd hour
  Measurements with Visual Analog Scale. Minimum value 0, maximum is 10. 0 is no pain and 10 is intolerable pain.
Postoperative Pain | Postoperatively 4th hour
  Measurements with Visual Analog Scale. Minimum value 0, maximum is 10. 0 is no pain and 10 is intolerable pain.
Postoperative Pain | Postoperatively 6th hour
  Measurements with Visual Analog Scale. Minimum value 0, maximum is 10. 0 is no pain and 10 is intolerable pain.
Postoperative Pain | Postoperatively 12th hour
  Measurements with Visual Analog Scale. Minimum value 0, maximum is 10. 0 is no pain and 10 is intolerable pain.
Postoperative Pain | Postoperatively 24th hour
  Measurements with Visual Analog Scale. Minimum value 0, maximum is 10. 0 is no pain and 10 is intolerable pain.

SECONDARY OUTCOMES:
Nausea and Vomiting | Postoperatively 5th minute
  Measurement with 4 point scale 0 no nausea
  1. mild nausea
  2. severe nausea
  3. vomiting
  4. severe and continuously vomiting
Nausea and Vomiting | Postoperatively 10th minute
  Measurement with 4 point scale 0 no nausea
  1. mild nausea
  2. severe nausea
  3. vomiting
  4. severe and continuously vomiting
Nausea and Vomiting | Postoperatively 15th minute
  Measurement with 4 point scale 0 no nausea
  1. mild nausea
  2. severe nausea
  3. vomiting
  4. severe and continuously vomiting
Nausea and Vomiting | Postoperatively 30th minute
  Measurement with 4 point scale 0 no nausea
  1. mild nausea
  2. severe nausea
  3. vomiting
  4. severe and continuously vomiting
Nausea and Vomiting | Postoperatively 60th minute
  Measurements with 4 point scale 0 no nausea
  1. mild nausea
  2. severe nausea
  3. vomiting
  4. severe and continuously vomiting
Nausea and Vomiting | Postoperatively 120th minute
  Measurements with 4 point scale 0 no nausea
  1. mild nausea
  2. severe nausea
  3. vomiting
  4. severe and continuously vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Yenimahalle, Turkey (Türkiye)